CLINICAL TRIAL: NCT05824871
Title: A Multicenter, Randomized, Double-Blind, Active-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Oral Sudapyridine (WX-081) Tablets in Patients With Rifampicin-Resistant Pulmonary Tuberculosis
Brief Title: A Phase III Study of Oral Sudapyridine (WX-081) Tablets in Rifampicin-Resistant Pulmonary Tuberculosis Patients
Acronym: WISH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JYP0081M301
Record Dates: First submitted 2023-04-10; First posted 2023-04-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-11

CONDITIONS: Rifampin-Resistant Pulmonary Tuberculosis; Tuberculosis, Multidrug-Resistant (MDR-TB)
Keywords: Rifampin-Resistant Tuberculosis; Multidrug-Resistant Tuberculosis (MDR-TB); Pulmonary Tuberculosis; Sudapyridine (WX-081); Bedaquiline; Antitubercular Agents; Randomized Controlled Trial; Background Regimen Therapy
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant; Tuberculosis, Pulmonary | interventions — sudapyridine; bedaquiline

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two groups (Sudapyridine and Bedaquiline) for parallel treatment evaluation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcome assessors will be blinded to the intervention assignments to ensure unbiased assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sudapyridine (WX-081) Group (Experimental): Participants in this group will receive Sudapyridine (WX-081) combined with background regimen (BR). Treatment starts with a loading dose of Sudapyridine for 2 weeks (450 mg once daily for 7 days, followed by 300 mg once daily for 7 days). This is followed by a maintenance dose of 150 mg once daily from Week 3 to Week 24. During the 24-week treatment period, participants will also receive a placebo for bedaquiline and continue their background regimen (BR). After the 24-week treatment period, participants will enter the background regimen phase and continue BR until Week 72.
  Interventions: Drug: Sudapyridine
- Bedaquiline Group (Active Comparator): Participants in this group will receive Bedaquiline combined with background regimen (BR). Treatment starts with a loading dose of Bedaquiline for 2 weeks (400 mg once daily), followed by a maintenance dose of 200 mg three times per week (with at least 48 hours between doses) from Week 3 to Week 24. During the 24-week treatment period, participants will also receive a placebo for Sudapyridine and continue their background regimen (BR). After the 24-week treatment period, participants will enter the background regimen phase and continue BR until Week 72.
  Interventions: Drug: Bedaquiline

INTERVENTIONS:
Drug: Sudapyridine — Sudapyridine (WX-081) will be administered as a loading dose for 2 weeks (450 mg once daily for 7 days, followed by 300 mg once daily for 7 days) and a maintenance dose (150 mg once daily) from Week 3 to Week 24. The intervention is combined with background regimen (BR) and placebo for bedaquiline.
  Other Names: WX-081
  Arms: Sudapyridine (WX-081) Group
Drug: Bedaquiline — Bedaquiline will be administered as a loading dose for 2 weeks (400 mg once daily) and a maintenance dose (200 mg three times per week, with at least 48 hours between doses) from Week 3 to Week 24. The intervention is combined with background regimen (BR) and placebo for Sudapyridine.
  Arms: Bedaquiline Group

SUMMARY:
This is a multicenter, randomized, double-blind, active-controlled Phase III study to evaluate the efficacy and safety of Sudapyridine (WX-081) combined with a background regimen (BR) in patients with rifampicin-resistant pulmonary tuberculosis.

Approximately 450 participants will be screened over a period of up to 2 weeks and randomized in a 2:1 ratio to receive either Sudapyridine or bedaquiline, in combination with placebo tablets and BR, for 24 weeks. After the treatment period, participants will enter a background regimen period up to Week 72, during which they will continue to receive BR.

A subset of participants will be included in the C-QT sub-study to assess intensive PK sampling and 12-lead ECG evaluations on Day 1 pre-dose, Day 14, and Week 24.

The study aims to provide robust data to support the use of Sudapyridine as a treatment option for rifampicin-resistant pulmonary tuberculosis.

DETAILED DESCRIPTION:
This Phase III clinical study is designed to evaluate the efficacy and safety of Sudapyridine (WX-081) in combination with a background regimen (BR) for the treatment of rifampicin-resistant pulmonary tuberculosis. The study will be conducted at multiple centers, employing a randomized, double-blind, active-controlled design.

The study will consist of three phases:

Screening Phase:

Duration: Up to 2 weeks. Approximately 450 participants with rifampicin-resistant pulmonary tuberculosis will be screened for eligibility.

Treatment Phase:

Participants will be randomized in a 2:1 ratio into two groups:

1. Sudapyridine Group: Sudapyridine (WX-081) with placebo and BR.
2. Bedaquiline Group: Bedaquiline with placebo and BR. Treatment duration: 24 weeks.

Background Regimen Phase:

After completing the treatment phase, participants in both groups will continue to receive the background regimen (BR) until Week 72.

The study aims to test the hypothesis that Sudapyridine (WX-081), when combined with a background regimen, is effective and safe for treating rifampicin-resistant pulmonary tuberculosis. The data collected from this study will include primary and secondary endpoints related to efficacy and safety, PK/PD data, and cardiac safety evaluations.

The sample size of approximately 450 participants is designed to provide adequate power to detect a statistically significant difference in outcomes between treatment groups. Comprehensive data validation procedures and a robust statistical analysis plan will ensure the reliability and accuracy of the results.

ELIGIBILITY:
Inclusion Criteria:

* • Body mass index (BMI) and body weight of subjects: 15.0≤BMI≤28.0 kg/m2, and 40kg≤ body weight ≤90kg;

  * For clinically diagnosed patients with tuberculosis whose drug sensitivity test has proved to be at least resistant to rifampicin, phenotypic or molecular drug sensitivity test results within 3 months before the subject signs informed consent can be accepted;
  * Direct sputum smear positive for acid-fast bacilli (AFB at least 1+);
  * Willing to discontinue all previous anti-tuberculosis drugs and accept a 7-day washout period;
  * Non-lactating and pregnant women who agree to use contraception throughout the treatment; Or the male patient's spouse agrees to use contraception throughout the treatment.

Exclusion Criteria:

* • Allergic to any study drug or its ingredients;

  * A history of alcohol dependence or drug abuse;
  * With hematogenous disseminated pulmonary tuberculosis or extrapulmonary tuberculosis;
  * Drug susceptibility test before screening showed resistance to more than 4 of the 8 antituberculosis drugs in this study;
  * Have taken Bedaquiline before;
  * HIV-positive patients;
  * Laboratory obvious abnormalities;
  * A history of pointy torsion ventricular tachycardia or cardiac risk factors for pointy torsion ventricular tachycardia;
  * Repeated QTcF intervals > 450ms; Clinically significant ventricular arrhythmias that may require medical or surgical treatment;
  * Documented cardiovascular diseases;
  * Peripheral neuropathy CTCAE grade 3 or grade 4; Grade 1 or grade 2 neuropathy that the investigator believes is likely to progress/worsen over the course of the study; optic neuritis;
  * Any serious cardiovascular, kidney, liver, blood, tumor, endocrine and metabolic, autoimmune or rheumatic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-10-22 (Estimated)

PRIMARY OUTCOMES:
Sputum Culture Conversion Rate at Week 24 | Week 24
  Proportion of participants achieving sputum culture conversion (SCC) at Week 24 of treatment, measured as a percentage.

SECONDARY OUTCOMES:
Time to Sputum Culture Conversion | Up to Week 72
  Time required for participants to achieve sputum culture conversion (SCC) during the study period.
Treatment Success Rate at Week 72 | Week 72
  Proportion of participants achieving treatment success at Week 72, based on predefined criteria.
Sputum Culture Conversion Rates at Multiple Time Points | Up to Week 72
  Proportion of participants achieving sputum culture conversion at Weeks 8, 12, 16, 20, 36, 48, 60, and 72.

CONTACTS AND LOCATIONS:
Overall Officials: Naihui Chu, Ph.D, Principal Investigator — Beijing Chest Hospital affiliated to Capital Medical University
Locations (2):
- China (2):
  - Beijing Chest Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No